CLINICAL TRIAL: NCT04999358
Title: The Effectiveness of a Targeted Protein Education Telehealth Intervention to Increase Protein Intake in Patients With Coronary Heart Disease and Low Protein Intake: A Pilot Study
Brief Title: Protein Intake in Patients With Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Emily James, Principal Investigator, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 296288
Record Dates: First submitted 2021-07-29; First posted 2021-08-10 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Coronary Heart Disease; Low Protein Intake; Sarcopenia
Keywords: Protein; Coronary heart disease; Rehabilitation; Telehealth
MeSH Terms: conditions — Coronary Disease; Sarcopenia

STUDY DESIGN:
Intervention Model Description: This is a single centre, parallel-group, two arm, randomised controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein group (Experimental): Participants in the protein group will receive their usual education session(s) as part of standard practice cardiac rehabilitation. The session(s) will be the same for both study arms and will align with the dietary education sessions that these patients would usually be given during their normal cardiac rehabilitation programme. Participants in the protein group will be provided with an additional targeted protein education session, which will aim to increase the amount of foods eaten with protein in them (≥1.2 g/kg protein/day) and improve the quality of protein sources that are eaten. The content and materials for these sessions can be provided in-person or are available as pre-recorded videos, accessed by participants via the internet or DVD
  Interventions: Behavioral: Protein education
- Control group (Placebo Comparator): Participants in the control group will receive their usual education session(s) as part of standard practice cardiac rehabilitation. The session(s) will be the same for both study arms and will align with the dietary education sessions that these patients would usually be given during their normal cardiac rehabilitation programme. Participants in the control group will receive an additional dietary education session that is similar to the standard practice sessions, containing only information that is usually provided in the cardiac rehabilitation programme.The content and materials for these sessions can be provided in-person or are available as pre-recorded videos, accessed by participants via the internet or DVD.
  Interventions: Behavioral: Standard education

INTERVENTIONS:
Behavioral: Protein education — The protein education session is pre-recorded and will describe in lay terms: the health issues associated with low protein intake, the amount of protein to eat in a day, and provide useful information to increase protein intake. This information will focus on the quality and amount of protein eaten, primarily using a whole-food approach. For example, the education sessions will give ideas for everyday foods that can be added to regular meals, favouring plant proteins, fish, lean meat, poultry, low fat dairy and eggs. The education session has been provided in conjunction with an NHS dietitian.
  Arms: Protein group
Behavioral: Standard education — Dietary advice provided as part of standard cardiac rehabilitation will be pre-recorded and provided to the control group. This education session will be in addition to usual care.
  Arms: Control group

SUMMARY:
Sarcopenia is a skeletal muscle disease, characterised by low muscle strength and muscle mass, and associated with higher medical care costs, shorter life expectancy and physical dependence. Sarcopenia affects around 1 in 10 older adults in the general population. However, in patients with coronary heart disease (CHD), this number is almost 3 in 10. Patients who have CHD are offered cardiac rehabilitation (CR); a multicomponent programme designed to improve long-term health outcomes. Nutritional education is an important part of CR and typically focuses around modifying fat and carbohydrate intake to lower cholesterol levels and achieve a healthy weight. Currently there is little focus on increasing protein intake, which might reduce the risk of sarcopenia. Eligible patients with CHD and low protein intake will receive the standard nutritional education delivered during CR. Next, participants will be randomised to one of two groups: protein education (intervention), or standard information (control). Whilst COVID-19 restrictions are in place, education will be delivered remotely via pre-recorded video. Outcome measures, including protein intake, sit to stand performance, sarcopenia risk score (modified SARC-F), Physical Activity Vital Signs (PAVS) and waist circumference, will be assessed at baseline, at the end of the standard CR programme and after a follow-up period of the same duration as the CR programme.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older.
* Recent diagnosis of coronary heart disease or a cardiac event related to coronary heart disease.
* Have been offered standard cardiac rehabilitation in a Newcastle upon Tyne Hospitals NHS Foundation Trust.
* Usually receive dietary education as part of their cardiac rehabilitation program.
* Able to understand and undertake the tasks described as part of this study.
* Able to provide written informed consent.

Exclusion Criteria:

* Patients advised against participation in light exercise by a medical professional.
* Patients younger than 50 years.
* Patients unable to alter their diet due to medical reasons; including patients that have been prescribed artificial feeding, texture modified diets, and specialist renal diets.
* Patients with known stage 4 or 5 chronic kidney disease.
* Patients without access to teleconferencing technology or without another adult present (≥18 years; and with capacity to supervise the activity) will be excluded from participating in the remote sit-to-stand test for their safety.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Change in protein intake (g/kg/day). | Up to 12 weeks and up to 24 weeks; time points determined by CR standard duration.
  Between-group intervention effect for dietary protein intake in the intervention and control groups. Protein intake is assessed with a three-day food diary.

SECONDARY OUTCOMES:
Prevalence of low protein intake in patients with coronary heart disease. | Baseline, up to 12 weeks and up to 24 weeks; time points determined by CR standard duration.
  Average protein intake and percentage of participants with protein intake <1.2 g/kg/day and <0.8 g/kg/day.
Change in sit to stand performance (leg strength). | Up to 12 weeks and up to 24 weeks; time points determined by CR standard duration.
  Between-group intervention effect for sit to stand performance in the intervention and control groups. The time taken to complete five consecutive sit to stands will be recorded.
Change in sarcopenia risk score and self-reported physical activity. | Up to 12 weeks and up to 24 weeks; time points determined by CR standard duration.
  Between-group intervention effect for questionnaire scores in the intervention and control groups. Sarcopenia risk and physical activity are assessed using the modified SARC-F questionnaire (SARC-F+EBM; includes age and body mass index) and Physical Activity Vital Signs questionnaire (PAVS), respectively.
Difference in protein intake between patients with and without probable sarcopenia. | Baseline, up to 12 weeks and up to 24 weeks; time points determined by CR standard duration.
  Probable sarcopenia is assessed using sit to stand time. The cut-off point for probable sarcopenia will be >15seconds to complete five sit to stands, as proposed by the European Working Group on Sarcopenia in Older People-2.
Change in waist circumference. | Up to 12 weeks and up to 24 weeks; time points determined by CR standard duration.
  Between-group intervention effect for waist circumference will be assessed as a simple indicator of body composition.
Reliability of self-assessed waist circumference. | 24 hours.
  Whilst COVID-19 restrictions are in place, participants will be required to complete their own waist circumference measurement. Measures will be taken 24 hours apart to determine their reliability.
Adherence | Up to 12 weeks.
  Adherence will be assessed as the amount of education sessions completed by participants, as a percentage of those prescribed.
Attrition. | Up to 12 weeks and up to 24 weeks; time points determined by CR standard duration.
  Attrition will be assessed as the percentage of participants that drop out of the intervention before the study period is complete.
Occurrence of adverse events | Up to 12 weeks and up to 24 weeks; time points determined by CR standard duration.
  Adverse events (such as injury or illness) that are directly related to the intervention will be reported..
Understanding and evaluation of the intervention. | Baseline and up to 12 weeks.
  A short questionnaire will determine patients' understanding of the educational material and their evaluation of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair O'Doherty, PhD, Study Chair — University of Northumbria at Newcastle
Locations (1):
- Newcastle upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No